CLINICAL TRIAL: NCT02929836
Title: Optimal Ablation Endpoint for Longstanding Persistent Atrial Fibrillation: a Randomized Prospective Study
Brief Title: Catheter Ablation of Longstanding Persistent Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, wang yuanlong, MD, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DSL-20161002
Record Dates: First submitted 2016-10-05; First posted 2016-10-11 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Atrial Fibrillation
Keywords: Ablation Linear Lesions
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PVI+LA linear ablation +CFAE ablation (Active Comparator): The ablation procedure for atrial fibrillation guided by CARTO system, including PVI, LA linear ablation (roof line and mitral isthmus)and CFAE ablation.
  Interventions: Procedure: PVI; Procedure: LA linear ablation; Procedure: CFAE ablation; Device: CARTO
- PVI+linear ablation +CFAE ablation (Active Comparator): The ablation procedure for atrial fibrillation guided by CARTO system, including PVI,roof line and mitral isthmus,cavotricuspid isthmus abaltion and CFAE ablation.
  Interventions: Procedure: PVI; Procedure: LA linear ablation; Procedure: CFAE ablation; Procedure: linear ablation; Device: CARTO
- PVI+CFAE ablation (Active Comparator): The ablation procedure for atrial fibrillation guided by CARTO system, including PVI and CFAE ablation.
  Interventions: Procedure: PVI; Procedure: CFAE ablation; Device: CARTO

INTERVENTIONS:
Procedure: PVI — PVI was the complete isolation of all PVs, which was confirmed by entrance and/or exit block into or from the PV antra.
Procedure: LA linear ablation — LA linear ablation include mitral isthmus ablation and roof line ablation. Mitral isthmus ablation (from the mitral annulus to the left inferior PV) was performed first, followed by roof line ablation (between the right and left superior PVs).
  Arms: PVI+LA linear ablation +CFAE ablation; PVI+linear ablation +CFAE ablation
Procedure: CFAE ablation — Ablation catheter was maintained in a stable position when the electrograms were being recorded for at least 5 s to avoid artifacts.The procedural endpoint of CFAEs was the complete elimination of fragmented atrial activity in local electrograms.
Procedure: linear ablation — Right atrial CTI ablation was performed during SR.
  Arms: PVI+linear ablation +CFAE ablation
Device: CARTO — 3 dimensional mapping system

SUMMARY:
This randomized prospective study compared three ablation strategies in patients with longstanding persistent atrial fibrillation (LPeAF). It also explored the best procedural endpoint from among the following: circumferential pulmonary vein isolation (PVI)+left atrial (LA) linear lesions (roof line, mitral isthmus)+complex fractionated atrial electrogram (CFAE) ablation, PVI+LA linear lesions +cavotricuspid isthmus (CTI) ablation +CFAE ablation, and PVI+CFAE ablation.

DETAILED DESCRIPTION:
Patients were randomized into three ablation groups: group A (n=100): PVI+LA linear ablation (roof line and mitral isthmus) +CFAE ablation; group B (n=100): PVI+linear ablation (roof line, mitral isthmus, and CTI) +CFAE ablation; group C (n=100), PVI+CFAE ablation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with longstanding persistent atrial fibrillation (lasting for>1 year)
* Exhibited refractoriness to at least one antiarrhythmic drug
* Left atrial diameter <=60mm

Exclusion Criteria:

* Patients with uncontrolled congestive heart failure
* Having significant valvular disease and/or prosthetic heart valve(s)
* With myocardial infarction or stroke within 6 months of screening
* With Significant congenital heart disease;ejection fraction was <40% measured by echocardiography
* Allergic to contrast media
* Contraindication to warfarin or heparin
* Severe pulmonary disease e.g. restrictive pulmonary disease
* Chronic obstructive disease (COPD)
* Left atrial (LA) thrombus measured by pre-procedure transesophageal echocardiography
* Having any contraindication to right or left sided heart catheterization
* Poor general health
* Life expectancy less than 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Time to first documented recurrence of atrial arrhythmias | 2-year follow-up
  Time to first documented recurrence of atrial arrhythmias after the first ablation procedure and after the final ablation procedure

SECONDARY OUTCOMES:
Procedure duration at ablation | At the end of the first ablation procedure
  Minutes elapsed from the first puncture of the femoral vein to the removal of the last catheter
Ablation time at ablation | At the end of the first ablation procedure ]
  Minutes elapsed from the onset of the first energy delivery to the end of the last energy delivery
Fluoroscopy time at ablation | At the end of the first ablation procedure
  Minutes of fluoroscopy used during the entire ablation procedure
Complications | 2-year follow-up
  Incidence of peri-procedural complications including stroke, PV stenosis, cardiac perforation, esophageal injury, and death.
Type of recurrent arrhythmia | 2-year follow-up
  Specific type of recurrent atrial arrhythmia
Number of redo procedures | 2-year follow-up
  Number of redo procedures，including two or more procedures

CONTACTS AND LOCATIONS:
Overall Officials: Xu Mr Liu, MD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai chest hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No